CLINICAL TRIAL: NCT04487483
Title: Exploring the Impact of a Sleep App on Sleep Quality: a Randomised Controlled Pilot Study
Brief Title: Exploring the Impact of a Sleep App on Sleep Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Abi Fisher, Associate Professor of Physical Activity and Health, University College, London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SleepAppEvaluation
Record Dates: First submitted 2020-07-07; First posted 2020-07-27 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: The study is a two-arm pilot RCT where participants are randomly assigned to either the intervention or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep App (Experimental): Participants in this condition will receive full free access to the "Pro" version of the sleep app and asked to use the app every day for three months.
  Interventions: Behavioral: Sleep App
- Control (No Intervention): Participants in this condition will be asked to continue their life as normal and abstain from downloading or using any sleep aid and/or sleep tracker app for three months.

INTERVENTIONS:
Behavioral: Sleep App — A sleep app offering 6 evidence based techniques to improve sleep (such as Cognitive Behavioural Therapy for Insomnia, Progressive Muscle Relaxation and Mindfulness Meditation), allowing for a personally tailored journey of sleep aids within the app.
  Arms: Sleep App

SUMMARY:
Sufficient sleep is crucial for good health, yet a third of UK adults have impaired sleep quality. Therefore, there is urgent need for population-level sleep interventions. However, many sleep interventions (such as Cognitive Behavioural Therapy for Insomnia) are resource intensive and not widely available. Research demonstrates that smartphone interventions are an effective way to reach the wider population. However, many commercially available smartphone sleep applications focus on one technique, and hence do not tailor to the diverse needs of individuals. A new sleep app offers six different techniques, allowing individuals to shape their own journey to improved sleep quality. The investigators aim to test the sleep app's efficacy and gather user experience data to allow app optimisation. The study is a two-arm pilot randomised control trial (RCT). After recruitment and screening, baseline measurements will be taken: subjective sleep quality data will be collected using the Insomnia Severity Index (ISI) and the Consensus Sleep Diary from all participants and objective accelerometry data via an Oura Ring (worn on finger for a week) on a subsample of participants. Participants will then be randomised to the intervention or control. Intervention participants will be given free use of the sleep app for 3 months. Controls will be informed that they will not receive access to the intervention and will be asked to abstain from using any other digital sleep-based intervention during the 3 months. All participants will be given the ISI after each month and will be given the Consensus Sleep Diary to fill out for one week again after 2 months. The planned Oura ring follow-up after 2 months for participants who wore the Oura ring at baseline has been cancelled due to COVID-19. User engagement will be assessed using the Digital Behaviour Change Intervention Engagement Scale. Telephone interviews will also be conducted with 20-30 participants to explore experience of using the app, how the comparison group felt about being allocated to the control group and how the COVID-19 pandemic may have affected their sleep and other measures of the study. Change in self-reported sleep will be the primary outcome and qualitative user data secondary. Appropriate tests (such as an ANOVA or linear regression controlling for baseline sleep and testing for effect of group when using continuous data) and thematic analysis of qualitative interview data will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Own a smartphone

Exclusion Criteria:

* Having a clinically diagnosed sleep disorder for which they are currently being treated
* Frequent use (once a week or more) of any sleep medication
* Enrolment on another sleep trial
* Being unwilling to cease usage of other sleep apps for the duration of the study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported sleep quality | Baseline/1 month/2 months/3 months
  Measured using the Insomnia Severity Index. The scores from the Insomnia Severity Index range from 0 to 28, where higher scores indicate worse sleep quality.

SECONDARY OUTCOMES:
Change in self-reported sleep | Baseline/2 months
  Measured using the Consensus Sleep Diary.
Engagement with the sleep app | Once a week for 3 months
  Participant's responses to the Digital Behaviour Change Intervention Engagement Scale (only applicable to participants in the intervention group). The scores from the Digital Behaviour Change Intervention Engagement Scale range from 8 to 56, where higher scores indicate higher engagement.
Telephone interview qualitative user data | Up to 6 months
  Participant's qualitative responses to telephone interview questions about their experience of using the sleep app, how the comparison group felt about being allocated to the control group, and how the COVID-19 pandemic may have affected their sleep and other measures of the study (on a subsample of 20-30 participants).

CONTACTS AND LOCATIONS:
Overall Officials: Abi Fisher, Principal Investigator — University College, London
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pilot study and the investigators plan to disseminate findings in a peer reviewed publication and a masters thesis.

REFERENCES:
- [Derived] Armitage BT, Potts HWW, Irwin MR, Fisher A. Exploring the Impact of a Sleep App on Sleep Quality in a General Population Sample: Pilot Randomized Controlled Trial. JMIR Form Res. 2024 Aug 13;8:e39554. doi: 10.2196/39554. PMID 39137016

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT04487483/SAP_001.pdf